CLINICAL TRIAL: NCT06001723
Title: A Feasibility Study to Determine Whether the Botanical Garden Become a Region of Forest Therapy for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Collaborators: Taiwan Forestry Research Institute (Unknown)
Responsible Party: Principal Investigator, Chung-Hua Hsu, director of the hospital, Taipei City Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: TCHIRB-11104010
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms; Cancer; Mental Health Disorder; Depression
Keywords: Forest therapy; Forest healing; Cancer Survivors; Mental Health Disorder
MeSH Terms: conditions — Neoplasms; Mental Disorders; Depression | interventions — Forest Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Forest Therapy (Experimental): This is a pretest-posttest designed experiment. A two-hour guided forest healing activity was used as an intervention method. For the purpose of comparison, an urban area adjacent to the Taipei Botanical Garden, specifically the Wanhua district, was selected. This choice ensures the exclusion of extensive green spaces commonly used for walking.
  Interventions: Behavioral: Forest Therapy

INTERVENTIONS:
Behavioral: Forest Therapy — Forest healing activities are guided by professionals, allowing participants to engage in a two-hour sensory experience within the forest environment. This includes activities such as stacking leaves and stones, closing their eyes to listen to sounds, engaging in physical stretches, blindfolded tree identification, connecting with tree companions, creating earth mandalas, and partaking in tea ceremonies and sharing insights.

SUMMARY:
The forest healing system is an important topic of alternative therapy in recent years. To investigates forest therapy's effectiveness in alleviating negative emotions among post-cancer patients. It compares therapy outcomes at Taipei Botanical Garden and Fushan Botanical Garden. Utilizing a pretest-posttest experimental design, a two-hour guided forest healing activity serves as the intervention method. Data collection involves instrumental tests and saliva samples.

DETAILED DESCRIPTION:
Introduction:

Cancer's global impact persists, ranking among the top three causes of death in Taiwan. Despite improved survival rates after cancer surgery, negative emotions among patients remain a challenge. Post-cancer depression adversely affects treatment outcomes and overall quality of life. Forest therapy, a natural healing approach, has gained attention for its potential to reduce stress, mitigate negative emotions, and enhance well-being.

Objectives:

This study investigates forest therapy's effectiveness in alleviating negative emotions among post-cancer patients. It compares therapy outcomes at Taipei Botanical Garden and Fushan Botanical Garden. Additionally, the study explores the lasting emotional benefits of forest therapy.

Methods:

Utilizing a pretest-posttest experimental design, this study is conducted at the Botanical Garden in Fushan, Taipei. Participants are cancer patients who are six months post-treatment. A two-hour guided forest healing activity serves as the intervention method. Data collection involves instrumental tests and saliva samples. A comparable location adjacent to Taipei Botanical Garden, excluding urban areas, is selected for comparison activities. Portable heart rhythm monitors track data, and saliva samples are analyzed for salivary α-amylase enzyme kinetics and cortisol concentrations. The study employs questionnaires including the Profile of Mood States 2nd Edition-Adult short (POMS2-A short), Beck Depression Inventory-Second edition (BDI-II), Beck Anxiety Inventory (BAI), and the abbreviated Taiwan version of the World Health Organization Quality of Life-Brief (WHOQOL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* Over 20 year-old
* Cancer patients finished cancer treatments more than 6 months (regardless hormone therapy)
* Voluntary attendance

Exclusion Criteria:

* People who unable to walk for at least 120 minutes
* People who still smoking, chewing betel nut or drinking alcohol (over five standard cups in any situation)
* People who addicted to medicine
* People who attend another clinical trial at the same time or in the follow-up period of an interventional trial
* Pregnant women or breast feeding
* Other conditions that participants unable to cooperate with

Ages: 36 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
questionnaire: POMS2-A short (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of the Profile of Mood States 2nd Edition-Adult short at Fushan botanical garden
questionnaire: POMS2-A short (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of the Profile of Mood States 2nd Edition-Adult short at Taipei botanical garden
questionnaire: POMS2-A short (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of the Profile of Mood States 2nd Edition-Adult short at urban region
questionnaire: BAI (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of The Beck Anxiety Inventory at Fushan botanical garden
questionnaire: BAI (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of The Beck Anxiety Inventory at Taipei botanical garden
questionnaire: BAI (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of The Beck Anxiety Inventory at urban region
questionnaire: BDI-II (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of The Beck Depression Inventory II at Fushan botanical garden
questionnaire: BDI-II (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of baseline The Beck Depression Inventory II at Taipei botanical garden
questionnaire: BDI-II (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of baseline The Beck Depression Inventory II at urban region
questionnaire: WHOQOL-BREF (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of World Health Organization Quality of Life-Brief (Taiwan version) at Fushan botanical garden
questionnaire: WHOQOL-BREF (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of World Health Organization Quality of Life-Brief (Taiwan version) at Taipei botanical garden
questionnaire: WHOQOL-BREF (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of World Health Organization Quality of Life-Brief (Taiwan version) at urban region
physiological indicator: alpha-amylase activity in salivary (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of alpha-amylase activity in salivary by using commercial kits (Salimetrics®) at Fushan botanical garden
physiological indicator: alpha-amylase activity in salivary (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of alpha-amylase activity in salivary by using commercial kits (Salimetrics®) at Taipei botanical garden
physiological indicator: alpha-amylase activity in salivary (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of alpha-amylase activity in salivary by using commercial kits (Salimetrics®) at urban region
physiological indicator: cortisol concentration in salivary (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of cortisol concentration in salivary by using commercial kits (Salimetrics®) at Fushan botanical garden
physiological indicator: cortisol concentration in salivary (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of cortisol concentration in salivary by using commercial kits (Salimetrics®) at Taipei botanical garden
physiological indicator: cortisol concentration in salivary (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of cortisol concentration in salivary by using commercial kits (Salimetrics®) at urban region
physiological indicator: HRV (Heart Rate Variability) (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of HRV by using wrist monitors (ANSWatch®) to measure heart rate, heart rate variability (related to activities of the autonomic nervous system ANS), irregular heartbeats (IRRHB), and 5-minute continuous pulse wave at Fushan botanical garden
physiological indicator: HRV (Heart Rate Variability) (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of HRV by using wrist monitors (ANSWatch®) to measure heart rate, heart rate variability (related to activities of the autonomic nervous system ANS), irregular heartbeats (IRRHB), and 5-minute continuous pulse wave at Taipei botanical garden
physiological indicator: HRV (Heart Rate Variability) (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of HRV by using wrist monitors (ANSWatch®) to measure heart rate, heart rate variability (related to activities of the autonomic nervous system ANS), irregular heartbeats (IRRHB), and 5-minute continuous pulse wave at urban region
physiological indicator: blood pressures (systolic and diastolic) (Fushan botanical garden) | per-test → 2 hours intervention at Fushan botanical garden → post-test immediately after the intervention
  Change of blood pressures by using wrist monitors (ANSWatch®) to measure blood pressures (systolic and diastolic) at Fushan botanical garden
physiological indicator: blood pressures (systolic and diastolic) (Taipei botanical garden) | per-test → 2 hours intervention at Taipei botanical garden → post-test immediately after the intervention
  Change of blood pressures by using wrist monitors (ANSWatch®) to measure blood pressures (systolic and diastolic) at Taipei botanical garden
physiological indicator: blood pressures (systolic and diastolic) (urban region) | per-test → 2 hours intervention at urban region → post-test immediately after the intervention
  Change of blood pressures by using wrist monitors (ANSWatch®) to measure blood pressures (systolic and diastolic) at urban region

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD. PHD., Study Director — Branch of Chinese Medicine, Taipei City Hospital
Locations (1):
- Taipei city hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Wei RS, Chu YS, Hong MY, Li MY, Fan SW, Tung GS, Hsu CH. A comprehensive evaluation of the health benefits of forest therapy for cancer survivors. Environ Health Prev Med. 2026;31:7. doi: 10.1265/ehpm.25-00333. PMID 41605676